CLINICAL TRIAL: NCT05476393
Title: Comparison of Effectiveness of Erector Spinae Plane Block and Thoracal Paravertebral Block for Postoperative Analgesia After Cardiovascular Surgery: Randomized Study
Brief Title: ESPB vs TPVB for Cardiac Surgery
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: no participants
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Bahadir Ciftci, Primary researcher, Medipol University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Medipol Hospital 28
Record Dates: First submitted 2022-07-25; First posted 2022-07-27 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Cardiovascular Diseases
Keywords: Cardiovascular surgery; Postoperative pain management; Erector Spinae Plane Block; Thoracal paravertebral block
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Intervention Model Description: There are two models for this study. The first group is erector spinae plane block group. The second one is thoracal paravertebral block group.
Who Masked: Participant, Outcomes Assessor
Masking Description: The patient and the anesthesiologist who performs postoperative pain evaluation will not know the group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Erector spinae block (Group ESPB) (Active Comparator): ESP block will be applied in Group ESPB. The US probe will be placed longitudinally 2-3 cm lateral to the T5 transverse process. Three muscles from top to bottom; Trapezius at the top, rhomboid major in the middle, and the erector spina muscle at the bottom will be displayed over the hyperechoic transverse process. Using the in plane technique, the block needle will be advanced in the cranio-caudal direction and 5 ml of saline will be injected under the erector spina muscle and the block location will be confirmed. After the block location is confirmed, 40 ml of 0.25% bupivacaine will be administered (20 ml in each side).
  Interventions: Other: Postoperative management
- Thoracal paravertebral block group (Group TPVB) (Active Comparator): After visualizing the T5 spinous process sagittally with the US probe, the probe will be placed 2-3 cm laterally. The ribs and transverse processes will be displayed as hyperechoic structures. Superiorly, the costotransverse ligament and anteriorly the pleura will be visualized. With the in-plane technique, the block needle will be advanced in the cranio-caudal direction until the costotransverse ligament is passed. 5 ml of saline will be injected and the block location will be confirmed. After confirming the location of the needle, negative aspiration is performed, and after observing the absence of CSF, blood and air, 40 ml of 0.25% bupivacaine will be administered, and it will be seen that the pleura is pushed down as the drug is administered (20 ml in each side).
  Interventions: Other: Postoperative management

INTERVENTIONS:
Other: Postoperative management — 1 g paracetamol will be administered 3 x 1. If the NRS score is ≥ 4, 1 mg kg-1 iv tramadol will be administrated.

SUMMARY:
Pain is a common and serious problem after cardiovascular surgery. It is associated with increased morbidity and mortality, and additional risk factors of cardiac surgery such as sternotomy and cardiopulmonary bypass contribute to this. Patient-controlled analgesia with intravenous opioids is standard in many centers for the management of pain after cardiac surgery. However, intravenous opioids have a higher risk of nausea and vomiting and may delay weaning from mechanical ventilation compared to regional techniques. Elderly patients have a higher risk of opioid-related complications, and regional techniques can help reduce postoperative ventilation time and accelerate postoperative recovery, which will reduce the risk of atelectasis, especially in the elderly population. Thoracic paravertebral block (TPVB) is difficult to apply due to its anatomical proximity to important structures such as the pleura and central neuraxial system, and may cause complications such as pneumothorax and vascular injury. Analgesia management is very important in these patients, since insufficient analgesia may cause pulmonary complications such as atelectasis, pneumonia, and increased oxygen consumption in the postoperative period.

Erector spina plane (ESP) block performed with ultrasound (US) is a new interfacial plane block defined by Forero et al. in 2016. If the ESP block is applied at the T5 level, it provides thoracic analgesia, if it is applied at the T7-9 level, it provides analgesia in the abdominal region.

In this study, it is aimed to compare the effectiveness of US-guided ESP block and TPVB for postoperative analgesia management after cardiovascular surgery. Our primary aim is to compare postoperative pain scores (NRS), and our secondary aim is to evaluate rescue analgesia using, opioid-related side effects (allergic reaction, nausea, vomiting) and complications that may occur due to block (pneumothorax, hematoma).

DETAILED DESCRIPTION:
Pain is a common and serious problem after cardiovascular surgery. It is associated with increased morbidity and mortality, and additional risk factors of cardiac surgery such as sternotomy and cardiopulmonary bypass contribute to this. Patient-controlled analgesia with intravenous opioids is standard in many centers for the management of pain after cardiac surgery. However, intravenous opioids have a higher risk of nausea and vomiting and may delay weaning from mechanical ventilation compared to regional techniques. Elderly patients have a higher risk of opioid-related complications, and regional techniques can help reduce postoperative ventilation time and accelerate postoperative recovery, which will reduce the risk of atelectasis, especially in the elderly population. Thoracic paravertebral block (TPVB) is difficult to apply due to its anatomical proximity to important structures such as the pleura and central neuraxial system, and may cause complications such as pneumothorax and vascular injury. Analgesia management is very important in these patients, since insufficient analgesia may cause pulmonary complications such as atelectasis, pneumonia, and increased oxygen consumption in the postoperative period.

Erector spina plane (ESP) block performed with ultrasound (US) is a new interfacial plane block defined by Forero et al. in 2016. If the ESP block is applied at the T5 level, it provides thoracic analgesia, if it is applied at the T7-9 level, it provides analgesia in the abdominal region. This block is applied by injecting a solution containing local anesthetic into the fascia under the erector spina muscle. Since the application site of the ESP block is far from the pleura and neuraxial tissues, it minimizes the risk of complications due to injury to these structures. Sonoanatomy is easy to visualize on US and the spread of local anesthetic can be seen easily. With the cephalo-caudal spread of the local anesthetic solution, analgesia occurs in several dermatomes. Cadaveric studies have shown that the injection spreads to the ventral and dorsal roots of the spinal nerves and creates sensory blockade in both the anterolateral thorax and the posterior. In the literature, it has been reported that it provides effective analgesia in randomized controlled studies investigating the effectiveness of ESP block for postoperative analgesia management after open heart surgery, breast surgery and ventral hernia repair.

In this study, it is aimed to compare the effectiveness of US-guided ESP block and TPVB for postoperative analgesia management after cardiovascular surgery. Our primary aim is to compare postoperative pain scores (NRS), and our secondary aim is to evaluate rescue analgesia using, opioid-related side effects (allergic reaction, nausea, vomiting) and complications that may occur due to block (pneumothorax, hematoma).

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) classification I-III
* Scheduled for cardiovascular surgery under general anesthesia

Exclusion Criteria:

* Bleeding diathesis
* anticoagulant treatment
* local anesthetics and opioid allergy
* Infection of the skin at the site of the needle puncture
* Patients who do not accept the procedure

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-08-30 (Actual); Primary Completion 2023-05-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain scores (Numerical Ratin Scala; 0=no pain, 10=the worst pain felt) | Postoperative 24 hours period
  Change from Baseline Pain Scores at Postoperative 24 hours.

SECONDARY OUTCOMES:
The need for rescue analgesia | Postoperative 24 hours period
  The amount of Tramodol using (mg)

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Medipol University Hospital, Istanbul, Bagcilar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared

REFERENCES:
- [Background] El Shora HA, El Beleehy AA, Abdelwahab AA, Ali GA, Omran TE, Hassan EA, Arafat AA. Bilateral Paravertebral Block versus Thoracic Epidural Analgesia for Pain Control Post-Cardiac Surgery: A Randomized Controlled Trial. Thorac Cardiovasc Surg. 2020 Aug;68(5):410-416. doi: 10.1055/s-0038-1668496. Epub 2018 Aug 16. PMID 30114712
- [Background] Nagaraja PS, Ragavendran S, Singh NG, Asai O, Bhavya G, Manjunath N, Rajesh K. Comparison of continuous thoracic epidural analgesia with bilateral erector spinae plane block for perioperative pain management in cardiac surgery. Ann Card Anaesth. 2018 Jul-Sep;21(3):323-327. doi: 10.4103/aca.ACA_16_18. PMID 30052229
- [Background] Forero M, Adhikary SD, Lopez H, Tsui C, Chin KJ. The Erector Spinae Plane Block: A Novel Analgesic Technique in Thoracic Neuropathic Pain. Reg Anesth Pain Med. 2016 Sep-Oct;41(5):621-7. doi: 10.1097/AAP.0000000000000451. PMID 27501016
- [Background] D'Ercole F, Arora H, Kumar PA. Paravertebral Block for Thoracic Surgery. J Cardiothorac Vasc Anesth. 2018 Apr;32(2):915-927. doi: 10.1053/j.jvca.2017.10.003. Epub 2017 Oct 4. PMID 29169795